CLINICAL TRIAL: NCT00478270
Title: An Open Label Study to Assess the Effect of Intravenous Loading Doses of Bondronat on Metastatic Bone Pain in Patients With Breast Cancer and Skeletal Metastases.
Brief Title: A Study of Loading Doses of Intravenous Bondronat (Ibandronate) in Patients With Breast Cancer and Metastatic Bone Disease.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20247
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Pain; Bone Neoplasm; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bondronat]

INTERVENTIONS:
Drug: ibandronate [Bondronat] — 6mg iv on days 1-3

SUMMARY:
This single arm study will assess the efficacy of loading doses of intravenous Bondronat in reducing pain in patients with breast cancer and metastatic bone disease experiencing moderate to severe bone pain. Patients will receive an intravenous infusion of 6mg Bondronat on days 1, 2 and 3. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* breast cancer;
* bone metastases;
* mean worst pain score >=4 during 3 day baseline period;
* stable dose of analgesics over a 3 day baseline period;
* adequate renal function.

Exclusion Criteria:

* bisphosphonate treatment within 3 weeks of study enrollment;
* a change in antineoplastic treatment within 6 weeks of study enrollment;
* bone radiation within 2 weeks of study enrollment;
* active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pain response (20% decrease in mean pain score compared to baseline, and <=50% increase in mean analgesic consumption | Days 5 - 7

SECONDARY OUTCOMES:
Mean worst pain score over first 7 days | Day 7
Analgesic consumption | Day 7
Karnofsky index | Day 7
AEs, laboratory parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Greece (6):
  - Alexandroupoli
  - Athens
  - Haidari
  - Pátrai
  - Piraeus
  - Thessaloniki